CLINICAL TRIAL: NCT04086277
Title: Continuous Intrapartum Support to Reduce Primary Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMSS Hospital General de Zona 4, Celaya, Guanajauto, Mexico (Other Government)
Collaborators: Fondo de Investigación en Salud (FIS), México (Unknown)
Responsible Party: Principal Investigator, Luz Maria Cardona Torres, Subjefe de Educación e Investigación en Salud, IMSS Hospital General de Zona 4, Celaya, Guanajauto, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LMCT-02
Record Dates: First submitted 2019-09-06; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; Continuous intrapartum support; nulliparous

STUDY DESIGN:
Intervention Model Description: The control group was composed of women with labour, who attended the General Hospital of Zone 4 of the Guanajuato Delegation of the IMSS in the period of October-December 2016. The study group was composed of women with labour who presented at the same hospital to receive obstetric care in the period of October - December 2018.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women in labor with continuous intrapartum support (Experimental): Continuous intrapartum support was based on three basic aspects: 1) emotional support, 2) physical support and comfort measures and 3) information and advice.
  Interventions: Procedure: Continuous Intrapartum Support
- Women in labor without continuous intrapartum support. (No Intervention): The no intervention group received the usual obstetric care, without continuous intrapartum support.

INTERVENTIONS:
Procedure: Continuous Intrapartum Support — Received the usual obstetric care plus continuous intrapartum support that was provided by a Bachelor of Nursing and Obstetrics who received prior training by a professional doula.
  Arms: Women in labor with continuous intrapartum support

SUMMARY:
The objective of the study was to evaluate the intervention of intrapartum continuous support by a professional nurse with a university degree to reduce the nulliparous, term, singleton, vertex (NTSV) cesarean birth rate, in women pregnant less than 40 years in the HGZ No. 4 of the Guanajuato delegation of the Mexican Institute of Social Security, Mexico

DETAILED DESCRIPTION:
Continuous intrapartum support is a strategy used to decrease the cesarean section rate, where multiple factors influence its effectiveness (start and duration of support, professional training of support staff, and others.). The objective of the study was to decrease the rate of deliveries by cesarean, through continuous intrapartum support during the active phase until birth, by a professional nurse with a university degree, the support was based on three basic aspects: 1) emotional support, 2) physical support and comfort measures and 3) information and counseling, for which a quasi-experimental study was conducted, with a study population of 115 women in labour (nulliparous, full-term, single product, vertex position) and under 40 years, a group control was formed (n = 55) who received routine maternal care and a study group (n = 60) who received continuous intrapartum support.

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant
* Nulliparous
* Term pregnancy
* Singleton pregnancy
* Vertex position

Exclusion Criteria:

* Patients with maternal, fetal, or mixed cesarean indications were excluded.

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Cesarean delivery rate | Until the occurrence of delivery (expected range from 6 hours to 12 hours)
  Percentage de cesarean section in the arms

SECONDARY OUTCOMES:
Time of labour | From the active phase up to delivery (expected range from 6 hours to 12 hours)
  Labour covered the period of time from the active phase to birth. (Hours)
Apgar score | At 1 and 5 minutes after delivery
  Is a quick test performed on a baby at 1 and 5 minutes after birth
Obstetric analgesia | From the active phase up to delivery (expected range from 6 hours to 12 hours)
  If obstetric analgesia was applied to reduce the pain of labour. (Yes/No)
  If obstetric analgesia was applied to reduce the pain of labour. (Yes/No)
Induction of labour | start of active phase (up to 1 hour)
  If oxytocin was used to induce labour. (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Luz M Cardona, Master, Principal Investigator — IMSS Hospital General de Zona 4, Celaya, Guanajauto, México
Locations (1):
- IMSS Hospital General de Zona 4, Celaya, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Through a public web address
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since its publication, minimum 5 years.
Access Criteria: web address
URL: https://i0000.clarodrive.com/s/B87gCxXmS4DgyqK

REFERENCES:
- [Background] World Health Organization and Human Reproduction Programme. WHO Statement on Caesarean Section Rates. Statement. Geneva, Switzerland: World Health Organization, Department of Reproductive Health and Research ; 2015.
- [Background] Bohren MA, Hofmeyr GJ, Sakala C, Fukuzawa RK, Cuthbert A. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2017 Jul 6;7(7):CD003766. doi: 10.1002/14651858.CD003766.pub6. PMID 28681500
- [Background] Kabakian-Khasholian T, Portela A. Companion of choice at birth: factors affecting implementation. BMC Pregnancy Childbirth. 2017 Aug 31;17(1):265. doi: 10.1186/s12884-017-1447-9. PMID 28854903
- [Background] McGrath SK, Kennell JH. A randomized controlled trial of continuous labor support for middle-class couples: effect on cesarean delivery rates. Birth. 2008 Jun;35(2):92-7. doi: 10.1111/j.1523-536X.2008.00221.x. PMID 18507579
- [Background] Kashanian M, Javadi F, Haghighi MM. Effect of continuous support during labor on duration of labor and rate of cesarean delivery. Int J Gynaecol Obstet. 2010 Jun;109(3):198-200. doi: 10.1016/j.ijgo.2009.11.028. Epub 2010 Feb 12. PMID 20152972
- [Background] Khresheh R. Support in the first stage of labour from a female relative: the first step in improving the quality of maternity services. Midwifery. 2010 Dec;26(6):e21-4. doi: 10.1016/j.midw.2008.11.003. Epub 2009 Jan 6. PMID 19128863
- [Background] Wang M, Song Q, Xu J, Hu Z, Gong Y, Lee AC, Chen Q. Continuous support during labour in childbirth: a Cross-Sectional study in a university teaching hospital in Shanghai, China. BMC Pregnancy Childbirth. 2018 Dec 6;18(1):480. doi: 10.1186/s12884-018-2119-0. PMID 30522458